CLINICAL TRIAL: NCT00140608
Title: Efficacy of Seprapack Sinus Dressing Versus No Dressing in the Prevention of Intranasal Adhesions Following Sinus Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPACK00104ORP
Record Dates: First submitted 2005-08-29; First posted 2005-09-01 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Sinusitis
Keywords: sinus
MeSH Terms: conditions — Fistula

INTERVENTIONS:
Device: Seprapack Sinus Dressing

SUMMARY:
The purpose of this study is to investigate if the space occupying effect of Seprapack will lead to a reduction in post operative adhesions and more healing of the sinus cavity when compared to the use of no packing material.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* requiring bilateral endoscopic ethmoidectomy (anterior or posterior)
* intact middle turbinates
* willing to return for all follow-up visits
* signed written informed consent

Exclusion Criteria:

* patients with craniofacial abnormalities (e.g. cleft palate)
* patients without intact middle turbinates
* patients on long-term oral steroids or other chemotherapeutic agents that might delay healing. Short-term pulse steroid therapy and topical steroids are acceptable
* patients with inflammatory conditions, other than chronic sinusitis or nasal polyposis, including but not limited to sarcoidosis, rhinitis, ozena, Wegner's granulomatosis, nasal malignancy, recreational drug abuse
* patients with cystic fibrosis
* women that are pregnant or women of childbearing age potential who are not practicing an acceptable method of birth control
* patients with bleeding disorders or who are receiving anticoagulants
* patients that may require a Lothrop procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Study Completion 2005-05

PRIMARY OUTCOMES:
reduction in post-operative scarring when compared to use of no sinus packing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- United States (3):
  - Medical University of South Carolina, Charleston, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - UT Health Science Center, Memphis, Tennessee